CLINICAL TRIAL: NCT03883464
Title: Quality of Life Related to Digestive Symptoms After Cholecistectomy. Short Term Effects of a Low Fat Intake.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Lluis Oms Bernad, Principal Investigator, Consorci Sanitari de Terrassa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 02-16-102-028
Record Dates: First submitted 2019-03-11; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Dyspepsia; Postoperative Complications; Quality of Life
Keywords: Quality of live; Cholecystectomy; Low fat diet; Postoperative
MeSH Terms: conditions — Dyspepsia; Postoperative Complications | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Randomly assigned low fat versus balanced diet following cholecystectomy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low fat intake (Experimental): Patients who underwent cholecystectomy and were instructed to have a low fat diet.
  Interventions: Other: Diet
- Regular diet (No Intervention): Patients who underwent cholecystectomy and were instructed to have a regular diet.

INTERVENTIONS:
Other: Diet — Restriction in postoperative fat diet
  Arms: Low fat intake

SUMMARY:
Background and aims: A low-fat diet has been traditionally recommended after cholecystectomy although evidence is lacking. The main aim of the study is to assess either if digestive symptoms improve following the operation and if the restriction of fat in diet does influence these symptoms.

Methods: Symptoms have to be prospectively assessed by the GIQLI score (Gastrointestinal Quality of Life Index) at baseline, and one month after cholecystectomy. A low fat diet or equilibrated diet is randomly assigned to patientes distributed in two groups (N=80) candidates to gallbladder removal. Patients have to follow the prescribed diet and complet a questionnaire of symptoms (GIQLI Symptomantic score).

DETAILED DESCRIPTION:
Introduction The post-cholecystectomy syndrome includes a heterogeneous group of gastrointestinal symptoms presenting after cholecystectomy. However, the term is inaccurate as it is frequently used both for biliary and non-biliary disorders. Liver function and imaging tests are key to rule out biliary disorders such as choledocolithiasis, bile duct injuries or biliary leaks that may have a specific treatment.

Symptoms of non-biliary disorders may persist or arise the novo after surgery. Patients may refer a large variation of symptoms including upper abdominal pain, dyspepsia, diarrhoea, constipation, bloating, flatulence, heartburn or nausea. However, data on prevalence vary enormously. A recent systematic review underscored the lack of accurate data regarding post-cholecystectomy symptoms and only one of the 38 included studies fulfilled all quality criteria. This review showed a great variation of symptoms among the studies, diarrhoea being the most reported postoperative symptom but also with the largest variation across the studies. Moreover, the review found differences between persistent and de novo symptoms in the studies in which this distinction was made, showing that some symptoms considered to be due to the cholecystectomy may, however, be explained by coexisting pathologies such as irritable bowel syndrome or gastrointestinal disorders.

It has also been reported that most preoperative symptoms decrease after surgery except for diarrhoea, which may be a more persistent problem for a proportion of patients. However, data are controversial. Although some studies have reported a frequency of post-cholecystectomy diarrhoea between 5-12%, others support that new onset of diarrhoea is infrequent. A recent large population-based cohort study showed that cholecystectomy was associated with an increased risk of diarrhoea and stomach pain postoperatively, but a weakness of the study may be that questionnaires on gastrointestinal symptoms had not been validated.

Furthermore, a low-fat diet has been traditionally recommended after cholecystectomy for a variable period of time, but there is not a standard guideline on nutrition after surgery . Supposedly, the rationale for this recommendation is that the digestion of lipids may be hindered without the gallbladder. Other recommendations include a gradually increase of the fibre intake. However, literature addressing this issue is scarce and, to our knowledge, only three studies have assessed the effect of a low-fat diet on postoperative symptoms after cholecystectomy. One study failed to find differences in the postoperative symptoms between patients who followed a low-fat diet compared with a normal diet. On the contrary, two studies reported more postoperative symptoms in patients who did not follow a low-fat diet. The current situation is that there is a great variability in the dietary advice given by surgeons after surgery and, in addition, patients may or may not follow their recommendations making it more difficult to know whether specific dietary advice would be really necessary. A previous descriptive study carried by our group has evidenced the expected postoperative improvement in QoL and symtoms following the operation and has shown no differences in GIQLI scores between patients restricting fat intake and those following a diet without restriction.

Therefore, our aims is to prospectively assess symptoms after cholecystectomy by using a validated questionnaire and to assess the potential effect of the type of diet (fat restriction or banaced) followed after cholecystectomy.

Study design Prospective randomized trial in patients admitted at Consorci Sanitari de Terrassa (Barcelona, Spain) for treatment of symptomatic gallstone disease or its complications, evaluating short term postoperative digestive symptoms and if they are influenced by diet. Randomization according a random number table.

Group A: Low fat diet for hyperlipidemic conditions provided by Dietetics team. Group B: Balanced diet provided by Dietetics team

Participants Inclusion criteria: age > 18 years; symptomatic gallstone disease considering biliary pain or complications of gallstones (pancreatitis, cholangitis, cholecystitis).

Exclusion criteria: not willing to participate in the study, inability to understand the information due to mental disorders or language barrier; and severe postoperative complications which could affect the assessment of quality of life after cholecystectomy.

Assessments Prospective collection of patiens demographics, comorbidities and type of surgery. Score of digestive symptoms at baseline, and one month after the surgical procedure. Evaluations carried out during the visit at clinics at baseline and one month after surgery.

Completion the validated version of GIQLI score in Spanish, which has been widely used to assess the quality of life related to several digestive disorders including gallstone disease. The GIGLI is a 36-item patient reported outcomes instrument designed to assess GI-specific health-related quality of life and score from 0 to 4. Higher scores represent a better quality of life and the maximum score is 144. The GIGLI has five subscales: symptoms, physical function, emotional function, social function, and effects of treatment.

The symptoms subscale is the one considered in this study including:

Pain, Bloating, Epigastric fullness, Flatus, Belching, Abdominal noises, Bowel frequency, Restricted eating, Enjoyed eating, Regurgitation, Dysphagia, Eating speed, Nausea, Diarrhoea, Bowel urgency, Constipation, Blood in stod, Burning, Fecal incontinence.

Statistical analysis Descriptions of data will be presented as means and standard deviation for quantitative measures, and as absolute and relative frequencies for qualitative measures. Student's paired t test will be applied to assess differences in the GIGLI score between baseline and one month after treatment. Independent t-test will be applied to assess differences in the GIQLI overtime depending on the type of diet. A p-value <0.05 will be considered statistically significant. Sample size has been evaluated on the basis of standard deviation of the GIQLI score in our precedent descriptive study. Eighty patients per group for a beta error of 20% have to be included. Data analysis will be performed using the statistical Package SPSS version 20.

Ethical approval The study was approved by the Ethics Committees of the Consorci Sanitari de Terrassa. All patients provided written informed consent.

ELIGIBILITY:
Inclusion Criteria:

- Gallbladder removal because biliary pain or gallstones complications

Exclusion Criteria:

- Major postoperative complications, refusal to participate or not completion of questionnary.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Quality of Life (GIQLI)Symptoms | 1 month
  The Gastrointestinal Quality of Life Index (GIQLI) is a score validated in Spanish, that has been widely used to assess the quality of life related to several digestive disorders including gallstone disease. The GIGLI is a 36-item patient reported outcomes instrument designed to assess gastrointestinal quality of life. Items score from 0 to 4. Higher scores represent a better quality of life and the overall score ranges from 0 to 144, being a score 100 or higher indicative a good health status. This score has five subscales: symptoms, physical function, emotional function, social function, and effects of treatment.
  The symptoms subscale is the one considered and includes: Pain, Bloating, Epigastric fullness, Flatus, Belching, Abdominal noises, Bowel frequency, Restricted eating, Enjoyed eating, Regurgitation, Dysphagia, Eating speed, Nausea, Diarrhoea, Bowel urgency, Constipation, Blood in stod, Burning, Fecal incontinence. It scores from 0 to 76.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Oms, PhD, Principal Investigator — Consorci Sanitari de Terrassa; Luis Oms, PhD, Study Director — Consorci Sanitari de Terrassa
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Barcelona, Spain

REFERENCES:
- [Background] Plaisier PW. Cholecystectomy and bowel function. Gut. 2001 Feb;48(2):283. doi: 10.1136/gut.48.2.283. No abstract available. PMID 11211857
- [Background] Altomare DF, Rotelli MT, Palasciano N. Diet After Cholecystectomy. Curr Med Chem. 2019;26(19):3662-3665. doi: 10.2174/0929867324666170518100053. PMID 28521679
- [Background] Marcason W. What medical nutrition therapy guideline is recommended post-cholecystectomy? J Acad Nutr Diet. 2014 Jul;114(7):1136. doi: 10.1016/j.jand.2014.05.009. No abstract available. PMID 24956996
- [Background] Shin Y, Choi D, Lee KG, Choi HS, Park Y. Association between dietary intake and postlaparoscopic cholecystectomic symptoms in patients with gallbladder disease. Korean J Intern Med. 2018 Jul;33(4):829-836. doi: 10.3904/kjim.2016.223. Epub 2017 Nov 10. PMID 29117670
- [Background] Eypasch E, Williams JI, Wood-Dauphinee S, Ure BM, Schmulling C, Neugebauer E, Troidl H. Gastrointestinal Quality of Life Index: development, validation and application of a new instrument. Br J Surg. 1995 Feb;82(2):216-22. doi: 10.1002/bjs.1800820229. PMID 7749697
- [Background] Quintana JM, Cabriada J, Lopez de Tejada I, Varona M, Oribe V, Barrios B, Perdigo L, Bilbao A. Translation and validation of the gastrointestinal Quality of Life Index (GIQLI). Rev Esp Enferm Dig. 2001 Nov;93(11):693-706. English, Spanish. PMID 11995369
- [Background] Phillips SF. Diarrhea after cholecystectomy: if so, why? Gastroenterology. 1996 Sep;111(3):816-8. doi: 10.1053/gast.1996.v111.agast961110816. No abstract available. PMID 8780589
- [Background] Tan VP. The low-FODMAP diet in the management of functional dyspepsia in East and Southeast Asia. J Gastroenterol Hepatol. 2017 Mar;32 Suppl 1:46-52. doi: 10.1111/jgh.13697. PMID 28244670
- [Background] Khodarahmi M, Azadbakht L. Dietary fat intake and functional dyspepsia. Adv Biomed Res. 2016 Apr 21;5:76. doi: 10.4103/2277-9175.180988. eCollection 2016. PMID 27195249
- [Result] Jaunoo SS, Mohandas S, Almond LM. Postcholecystectomy syndrome (PCS). Int J Surg. 2010;8(1):15-7. doi: 10.1016/j.ijsu.2009.10.008. Epub 2009 Oct 24. PMID 19857610
- [Result] Filip M, Saftoiu A, Popescu C, Gheonea DI, Iordache S, Sandulescu L, Ciurea T. Postcholecystectomy syndrome - an algorithmic approach. J Gastrointestin Liver Dis. 2009 Mar;18(1):67-71. PMID 19337637
- [Result] Lublin M, Crawford DL, Hiatt JR, Phillips EH. Symptoms before and after laparoscopic cholecystectomy for gallstones. Am Surg. 2004 Oct;70(10):863-6. PMID 15529838
- [Result] Lamberts MP, Lugtenberg M, Rovers MM, Roukema AJ, Drenth JP, Westert GP, van Laarhoven CJ. Persistent and de novo symptoms after cholecystectomy: a systematic review of cholecystectomy effectiveness. Surg Endosc. 2013 Mar;27(3):709-18. doi: 10.1007/s00464-012-2516-9. Epub 2012 Oct 6. PMID 23052498
- [Result] Fort JM, Azpiroz F, Casellas F, Andreu J, Malagelada JR. Bowel habit after cholecystectomy: physiological changes and clinical implications. Gastroenterology. 1996 Sep;111(3):617-22. doi: 10.1053/gast.1996.v111.pm8780565.
- [Result] Ros E, Zambon D. Postcholecystectomy symptoms. A prospective study of gall stone patients before and two years after surgery. Gut. 1987 Nov;28(11):1500-4. doi: 10.1136/gut.28.11.1500. PMID 3428678
- [Result] Wilson RG, Macintyre IM. Symptomatic outcome after laparoscopic cholecystectomy. Br J Surg. 1993 Apr;80(4):439-41. doi: 10.1002/bjs.1800800410. PMID 8495304
- [Result] Sauter GH, Moussavian AC, Meyer G, Steitz HO, Parhofer KG, Jungst D. Bowel habits and bile acid malabsorption in the months after cholecystectomy. Am J Gastroenterol. 2002 Jul;97(7):1732-5. doi: 10.1111/j.1572-0241.2002.05779.x. PMID 12135027
- [Result] Luman W, Adams WH, Nixon SN, Mcintyre IM, Hamer-Hodges D, Wilson G, Palmer KR. Incidence of persistent symptoms after laparoscopic cholecystectomy: a prospective study. Gut. 1996 Dec;39(6):863-6. doi: 10.1136/gut.39.6.863. PMID 9038671
- [Result] Hearing SD, Thomas LA, Heaton KW, Hunt L. Effect of cholecystectomy on bowel function: a prospective, controlled study. Gut. 1999 Dec;45(6):889-94. doi: 10.1136/gut.45.6.889. PMID 10562588
- [Result] Talseth A, Edna TH, Hveem K, Lydersen S, Ness-Jensen E. Quality of life and psychological and gastrointestinal symptoms after cholecystectomy: a population-based cohort study. BMJ Open Gastroenterol. 2017 Apr 1;4(1):e000128. doi: 10.1136/bmjgast-2016-000128. eCollection 2017. PMID 28761686
- [Result] de Menezes HL, Fireman PA, Wanderley VE, de Menconca AM, Bispo RK, Reis MR. Randomized study for assessment of hypolipidic diet in digestive symptoms immediately following laparoscopic cholecystectomy. Rev Col Bras Cir. 2013 May-Jun;40(3):203-7. doi: 10.1590/s0100-69912013000300007. English, Portuguese. PMID 23912367
- [Result] Yueh TP, Chen FY, Lin TE, Chuang MT. Diarrhea after laparoscopic cholecystectomy: associated factors and predictors. Asian J Surg. 2014 Oct;37(4):171-7. doi: 10.1016/j.asjsur.2014.01.008. Epub 2014 Mar 17. PMID 24647139
- [Result] Lamberts MP, Den Oudsten BL, Keus F, De Vries J, van Laarhoven CJ, Westert GP, Drenth JP, Roukema JA. Patient-reported outcomes of symptomatic cholelithiasis patients following cholecystectomy after at least 5 years of follow-up: a long-term prospective cohort study. Surg Endosc. 2014 Dec;28(12):3443-50. doi: 10.1007/s00464-014-3619-2. Epub 2014 Jun 21. PMID 24950724